CLINICAL TRIAL: NCT06716047
Title: Effects of DL-endopeptidase Produced by Probiotics on Human Intestinal NOD2 Ligands and Related Functions
Brief Title: Effects of DL-endopeptidase Producing Probiotics on Human Intestinal NOD2 Ligands and Related Functions
Acronym: probiotics
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ZhujiangHZD
Record Dates: First submitted 2024-10-14; First posted 2024-12-04 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Microecological Therapy; Probiotic Intervention
Keywords: probiotics; safty; microecological therapy
MeSH Terms: interventions — Administration, Oral

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): resistant dextrin
  Interventions: Other: Oral administration
- probiotics (Experimental): lactobacillus
  Interventions: Other: Oral administration

INTERVENTIONS:
Other: Oral administration — Take it directly

SUMMARY:
We have discovered a type of probiotic that can target activating intestinal NOD2, which is related to a series of human health issues.

DETAILED DESCRIPTION:
This trial requires the subjects to take probiotics for a certain period of time, and we will collect blood, stool and questionnaires for subsequent testing, efficacy evaluation and safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Tend to participate the trial
* Willing to provide written informed consent

Exclusion Criteria:

* Recent use of probiotics, antibiotics, laxatives, or gastrointestinal ulcer medications within the past month.
* Gastrointestinal symptoms (e.g., constipation, abdominal pain, diarrhea, melena, hematochezia) in the past month.
* Other conditions considered by researchers for exclusion

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-12-05 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
safty | up to 2 weeks
  Adverse reaction by questionnaire survey
NOD2 activation level | up to 2 weeks
  the level of NOD2 activation by fecal in vitro experiments

SECONDARY OUTCOMES:
Intestinal barrier | up to 2 weeks
  Intestinal Barrier markers

CONTACTS AND LOCATIONS:
Locations (1):
- Industrial Avenue 253, canton, Guangzhou, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No
For personal privacy security